CLINICAL TRIAL: NCT03113149
Title: Which Factors Are the Strongest Predictors of a Positive Outcome After Physiotherapy for Patients With Knee Osteoarthritis?
Brief Title: Strongest Predictors of a Positive Outcome After Physiotherapy for Knee Osteoarthritis
Status: Terminated | Type: Observational
Why Stopped: Recruitment too slow, probably due to the procedure considered too complicated.
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University Hospital, Umeå (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/984-1
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Physical Therapy Modalities; Recovery of Function; Predictive Value of Tests; Cohort Studies
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- knee osteoarthritis: Patients with knee osteoarthritis after having started physical therapy

SUMMARY:
Individuals with painful knee osteoarthritis (OA) experience restricted physical function. Few previous studies have investigated comprehensive sets of constructs and tests to investigate physical function in these patients. Most single studies of knee OA patients show limited scope for explaining physical function in the perspective of WHO's International Classification of Functioning, Disability and Health (ICF) 3 levels: Body functions (the bodily level), Activities (individual level), and Participation (societal level). On the bodily level there is limited case-control knowledge on muscle strength beyond the knee and endurance-strength in general. On the activity level, there is similar limitation of biomechanical bodily features in stair climbing. On the participation level the situation is similar for objective performance. Measures are needed that inter-relate all three levels of ICF. These should also include well discriminating tests e.g. knee strength, walking, and activities of daily life (ADL), as well as both objective and subjective measures.

The purpose of this study is to explore mechanisms that can explain physical function in patients with knee OA in primary care. The study's main and primary goal is to quantify which baseline factors and change scores are the strongest predictors of a positive treatment outcome in terms of patients' global perceived change after physiotherapy. Secondary research question is: which factors are the strongest predictors of a positive outcome of physiotherapy in knee OA, in terms of pain intensity, patient specific functional scale, and function in daily living?

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and radiological osteoarthritis of the knee and referred to physiotherapists.
2. Symptomatic daily during the last month.
3. Symptomatic for more than one year.
4. Able to walk up and down a flight of 10 stairs with or without walking aids.
5. Able to walk 3 stairs up and down without walking aids.
6. Understand Norwegian orally and in writing.
7. Body mass index below 35.

Exclusion Criteria:

1. Neurological, rheumatic, orthopedic, or respiratory diagnosis, other than osteoarthritis of the knee which can negatively affect the walking ability, balance or pain.
2. Body mass index above or equal to 35.
3. Fracture of the femur or shank, or arthroscopic surgery in the osteoarthritic knee.
4. Chronic generalized pain (American College of Rheumatology Criteria, 2010).
5. Inability to understand Norwegian language.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee OA patients recruited from a private physiotherapy practice in Trondheim, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
patient global perceived effect | Change from baseline 'patient global perceived effect' at 3 months
  patient global perceived effect scale (Dworkin 2005, Evans 2014)

SECONDARY OUTCOMES:
Patient Specific Functional Scale | Change from baseline 'Patient Specific Functional Scale' at 3 months
  Patient Specific Functional Scale (Stratford, 1995)
Pain intensity | Change from baseline 'Pain intensity' at 3 months
  Pain Intensity scale (Dworkin 2005)
Function of daily living | Change from baseline 'Function of daily living' at 3 months
  Function of daily living scale (KOOS) (Roos & Lohmander 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuromedicine and Movement Science, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided